CLINICAL TRIAL: NCT03505697
Title: The Effects of Inspiratory Muscle Training on Exercise Capacity, Dyspnea and Lung Functions in Lung Transplantation Candidates
Brief Title: The Effects of IMT on Exercise Capacity, Dyspnea and Lung Functions in LTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: esrapehlivan
Record Dates: First submitted 2018-04-07; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Lung Transplant; Inspiratory Muscle Training
Keywords: rehabilitation; exercise; maximal inspiratory pressure; 6-minute walk test
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT+PR Group (Experimental): Patients received a 3-month standard hospital-based Pulmonary Rehabilitation included aerobic and strength training. In addition standard pulmonary rehabilitation, patients received inspiratory muscle training.
  Interventions: Other: inspiratory muscle training; Other: Pulmonary rehabilitation
- PR group (Experimental): Patients received a 3-month standard hospital-based Pulmonary Rehabilitation included aerobic and strength training.
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: inspiratory muscle training — Inspiratory Muscle Training was performed with an exercise tool (Powerbreath®) with a resistance range of 0-90. The training intensity was started with 30% of the Maximum Inspiratory Pressure (MIP) value obtained as a result of the mouth pressure measurement16, training was progressively increased from 30% to 60% considering that they were terminal-stage pulmonary disease patients. Patients were asked to perform IMT for 15 minutes, twice a day, 7 days a week, for 3 months.
  Arms: IMT+PR Group
Other: Pulmonary rehabilitation — Aerobic training:The aerobic exercise program consists of treadmill walking, cycle ergometer and arm ergometer training. Group exercises were performed in sets of 15 minutes each with three exercise modalities.
  Strength training:It is recommended that resistance targets are set at loads equivalent to 20 to 40% of a 1-repetition maximum (1RM) maneuver and performed between 8 to 12 repetitions for 1 to 2 sets per session.
  Home exercise programme:The program included breathing exercises (local expansion exercises, diaphragmatic breathing and pursed lip breathing), free walking, upper and lower extremity strengthening exercises with Thera-Band

SUMMARY:
Inspiratory Muscle Training (IMT), which is used to strengthen the respiratory muscles, is one of the techniques used in PR. It is mostly used in patients with chronic obstructive pulmonary disease, and has been shown to be beneficial for functionality and also for relieving dyspnea perception. It is reported in the guidelines that IMT has additional benefit for endurance in COPD patients. However, there are no studies related to its use and effectiveness in lung transplantation. In this study, we hoped to increase these known benefits by adding IMT to the standard Pulmonary Rehabilitation.

There are two main objectives of this study:

1. to examine the effect of respiratory muscle training on exercise capacity in lung transplantation candidates,
2. to compare dyspnea perception and lung function changes between the IMT+PR group and the PR group.

DETAILED DESCRIPTION:
The patients in the lung transplantation waiting list were included the study. These patients were with severe lung disease requiring transplantation, and that the intervention was undertaken before any lung transplantation. The patients were eligible for inclusion if they have: a diagnosis of terminally severe lung disease, being listed for lung transplantation, medically stable, had no orthopedic or cardiac problems that would prevent them from exercising and had no transfer problem to the PR centre.

Participants who meet the study inclusion criteria and complete the baseline assessments were randomly allocated into one of the two groups: namely Pulmonary Rehabilitation plus Inspiratory Muscle Training Group (IMT+PR) or Pulmonary Rehabilitation Group (PR) using a numbered series of 34 prefilled envelops specifying group assignment generated by a computer-based program.

All patients underwent supervised PR program on 2 days per week for 3 months. Apart from that, they were asked to perform the home exercise program which was scheduled as 3 days per week and fill out the exercise follow-up form. The study group was provided with IMT in addition to the standard program.

Statistical analysis was conducted using SPSS (version 15, USA). The Shapiro-Wilk statistic was used to test the normality of the distribution of all variables. Nonparametric tests were used in comparison, because the number of samples and the standard deviations of in-group chance (∆) were very large. The Wilcoxon Signed Rank Test was used to compare the pre- and post-treatment data of the groups, and the Mann-Whitney U test was used in the group-wise comparison. Nonparametric variables were expressed as median (minimum-maximum), and descriptive variables as percent. The chi-square test was used for categorical variables. Significance level was accepted as p <0.05 in all tests. We estimated that a sample size of 19 patients for each group to have 80% power with 5% type 1 error level to detect a minimum clinically significant differences of 54 meters of the 6-min walk test with the highest standard deviation of the study parameters.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of terminally severe lung disease,
* being listed for lung transplantation,
* medically stable,
* had no orthopedic or cardiac problems that would prevent them from exercising
* had no transfer problem to the PR centre.

Exclusion Criteria:

* Malignancy in the last 2 years,
* Other advanced major organ / system dysfunction that can not be treated outside the lung,
* Untreated non-pulmonary infection,
* Disputed medical treatment discontinuity,
* Untreatable psychiatric illness or psychosocial condition that interferes with treatment compliance,
* No appropriate, reliable social support,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Maximum Inspiratory Pressure (MIP) at 3-months | Three months
  The mouth pressure measurement was performed with the Micro-RPM® instrument from SensorMEDIC. Patient placed a rubber mouthpiece with flanges, on the device, sealed their lips firmly around the mouthpiece, exhaled/inhaled slowly and completely, and then tried to breath in as hard as possible. The patient was allowed to rest for about a minute and the maneuver was repeated five times. Verbal or visual feedback was provided after each maneuver. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value was obtained.
Change from baseline Maximum Expiratory Pressure (MEP) at 3-months | Three months
  The mouth pressure measurement was performed with the Micro-RPM® instrument from SensorMEDIC. Patient placed a rubber mouthpiece with flanges, on the device, sealed their lips firmly around the mouthpiece, exhaled/inhaled slowly and completely, and then tried to breath in as hard as possible. The patient was allowed to rest for about a minute and the maneuver was repeated five times. Verbal or visual feedback was provided after each maneuver. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value was obtained.
Change from baseline distance covered in six minute walking test at 3-months | Three months
  The test was conducted in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines. Patients were told that they should walk as fast as they can walk. Before and after the test, oxygen saturation, heart rate, Borg fatigue rating, and walking distance were recorded.
Change from baseline Modified Medical Research Council (mMRC) Dyspnea Scale score at 3-months | Three months
  Dyspnea perceptions during the activities of daily living were assessed with modified Medical Research Council (mMRC) scale.

SECONDARY OUTCOMES:
Change from baseline Forced Vital Capacity (FVC) at 3-months | Three months
  It was conducted by using the Sensor Medics model 2400 (Yorba Linda, CA, USA), and according to the American Thoracic Society (ATS) guidelines
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 3-months | Three months
  It was conducted by using the Sensor Medics model 2400 (Yorba Linda, CA, USA), and according to the American Thoracic Society (ATS) guidelines
Change from baseline alveolar volume ratio of carbonmonoxide diffusion capacity (DLCO/VA) at 3-months | Three months
  It was performed in the pulmonary function test laboratory using Cosmed Quark PFT (USA) with single breath technique

IPD SHARING:
Plan to Share IPD: No